CLINICAL TRIAL: NCT00692172
Title: An Open-Label, Multi-center Study to Evaluate the Safety and Tolerability of Intramuscular Administration of Alefacept (LFA-3/IgG1 Fusion Protein) in Subjects With Chronic Plaque Psoriasis Who Have Completed Studies C99-717 or C99-712
Brief Title: Open-label Study to Evaluate Safety of Multiple Courses of IM Alefacept During Treatment of Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-728
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Psoriasis
Keywords: psoriasis; alefacept; intramuscular
MeSH Terms: conditions — Psoriasis | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — intramuscular injection (IM)
  Other Names: Amevive; ASP0485

SUMMARY:
An extension study to evaluate safety and tolerability of up to 3 additional courses of IM alefacept in patients with chronic plaque psoriasis who have been previously treated with 1 or 2 courses of IM alefacept.

ELIGIBILITY:
Inclusion Criteria:

* Must have received at least 8 injections in the C99-717 study and completed the final follow-up visit OR,
* Must have completed the C99-712 study and been in C99-717 interim visits at the time dosing in the C99-717 study was closed. A subject who completed C99-712 but did not participate in any part of C99-717, including interim visits, must have prior sponsor approval before admission into C-728

Exclusion Criteria:

* Nursing mothers, pregnant women, and women planning to become pregnant while on study are to be excluded. Female patients who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study
* Clinically significant abnormal hematology values or history of an immunosuppressive disorder
* Serious local infection or systemic infection within 3 months prior to the first dose of alefacept
* A significant change in the subject's medical history from their previous alefacept study
* Any subject who initiated alternative systemic therapy, phototherapy, or disallowed therapy prior to visit 8 in study C99-712 or C99-717
* Current enrollment in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy (participation in registry-type studies is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2001-12; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety including evaluation of incidence of adverse events, physical exams and laboratory monitoring | Throughout treatment course

SECONDARY OUTCOMES:
Proportion of subjects who achieved "Almost Clear" or "Clear" by Physicians' Global Assessment | Every 2 weeks throughout treamtent course

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (43):
- United States (19):
  - Hot Springs, Arkansas
  - Fresno, California
  - La Jolla, California
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Pinellas Park, Florida
  - Newnan, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Clinton Township, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Johnston, Rhode Island
  - Goodlettsville, Tennessee
  - Austin, Texas
  - San Antonio, Texas
- Belgium (3):
  - Brussels
  - Edegem
  - Liège
- Canada (8):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - London, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Sainte-Foy, Quebec
- Copenhagen, Denmark
- France (5):
  - Besançon
  - Brest
  - Nice
  - Paris
  - Tours
- Germany (3):
  - Bochum
  - Dresden
  - Munich
- Amsterdam, Netherlands
- Spain (2):
  - Madrid
  - Valencia
- Liverpool, United Kingdom

REFERENCES:
- [Background] Roberts JL, Ortonne JP, Tan JK, Jaracz E, Frankel E; Alefacept Clinical Study Group. The safety profile and sustained remission associated with response to multiple courses of intramuscular alefacept for treatment of chronic plaque psoriasis. J Am Acad Dermatol. 2010 Jun;62(6):968-78. doi: 10.1016/j.jaad.2009.07.032. Epub 2010 Apr 14. PMID 20392521